CLINICAL TRIAL: NCT01496976
Title: Phase II Study of Ofatumumab in Combination With High Dose Methylprednisolone Followed by Ofatumumab and Lenalidomide Consolidative Therapy for the Treatment of Untreated CLL/SLL The HiLOG Trial
Brief Title: Ofatumumab, High Dose Methylprednisolone, Ofatumumab and Lenalidomide Consolidative Therapy for Untreated CLL/SLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16622; COMB157BUS21T (Other Grant/Funding Number: Novartis); RV-CLL-PI-0560 (Other Grant/Funding Number: Celgene Corp.)
Record Dates: First submitted 2011-12-16; First posted 2011-12-22 (Estimated); Results first posted 2021-12-02 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: leukemia; lymphoma; consolidative therapy; combination regimen; CLL; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Lymphoma | interventions — Methylprednisolone; ofatumumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immunotherapy (Experimental): Combination Regimen Followed by Consolidative Therapy: Ofatumumab/High Dose Methylprednisolone (HDMP) plus Ofatumumab/Lenalidomide
  Interventions: Drug: High Dose Methylprednisolone (HDMP); Drug: Ofatumumab; Drug: Lenalidomide

INTERVENTIONS:
Drug: High Dose Methylprednisolone (HDMP) — HDMP will be administered at 1 gm/m^2 IV over 90 minutes daily with ofatumumab infusions 1-8.
  Other Names: HDMP
Drug: Ofatumumab — Ofatumumab infusion will be administered immediately after HDMP.
  Other Names: Arzerra®
Drug: Lenalidomide — The Lenalidomide Starting Dose (Cycle 4) Based on Renal Function Prior to Cycle 4 of Treatment.
  Other Names: Revlimid®; IMiD® compound

SUMMARY:
The main purpose of this study is to see if ofatumumab with methylprednisolone followed by additional treatment with ofatumumab and lenalidomide can help people with Chronic Lymphocytic Leukemia (CLL) get rid of their CLL for a long period of time. Researchers also want to find out if the combination of ofatumumab with methylprednisolone followed by additional treatment with ofatumumab and lenalidomide is safe and tolerable.

DETAILED DESCRIPTION:
This is a phase II, single institution, and non-randomized study of patients with untreated CLL/SLL, utilizing a two-stage trial design. The primary endpoint for this trial is the combined complete and partial response rate (at 3 months-the end of cycle 3) to the protocol therapy. We anticipate this trial will have a complete response (CR) and partial response (PR) rate of at least 80%.

A two-stage design is employed for this trial. The null/unacceptable CR+PR response rate is ≤ 60% while the anticipated true response rate to the protocol treatment is at least 80% for each disease cohort. At the first stage, 26 patients will be accrued to the trial. If 15 or fewer of these patients respond, then the trial will be terminated early and the response rate to the protocol treatment will be deemed unacceptable (≤ 60%). Otherwise, if more than 15 patients respond during the first stage, an additional 19 patients will be enrolled to this trial during stage 2 for a total of 45 patients. If 32 or fewer of these 45 patients respond to the protocol treatment at the end of stage 2, no further investigation of the protocol treatment is considered warranted. On the other hand, if more than 32 patients out of the 45 enrolled patients respond, the protocol treatment will be considered promising. If the true response rate is ≤ 60%, the probability of ending the trial at stage 1 is 0.48. If, however, the true response rate is at least 80%, then the probability of ending the trial at stage 1 is only 0.01. This two-stage design has an overall alpha level of 0.045 and a power of 0.90.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Patients must have histologically or cytologically confirmed CD5+/CD20+ B-Cell chronic lymphocytic leukemia or small lymphocytic lymphoma. The diagnosis of CLL is based upon the National Comprehensive Cancer Network (NCCN) guidelines. Any outside pathology slides used as inclusion criteria for the patient will be reviewed at this institution to confirm the diagnosis. The patient must meet all of the following CLL criteria to participate in this study: absolute lymphocyte count > 5000/μL; CD20+ and CD5+; Bone marrow lymphocytes ≥ 30%; Or previous confirmed diagnosis of CLL/SLL with less than 5000/μl or less than 30% lymphocytes in bone marrow.
* Patients are eligible if they have stage III or IV disease. Patients with stage 0, I or II disease will be eligible if they have evidence of active disease defined as one or more of the following signs/symptoms: Documented weight loss of ≥ 10% over a 6 month period; Febrile episodes of 38 degrees Celsius (100.5 degrees F) or greater for greater than 2 weeks without evidence of infection; Massive or progressive splenomegaly defined as > 6 cm below the left costal margin; Massive (> 10 cm in longest diameter) or progressive lymphadenopathy.
* Patient has not received any prior treatment for CLL in the past.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 at study entry
* Laboratory test results within these ranges: Absolute neutrophil count ≥ 1000/mm³; Platelet count ≥ 50,000 /mm³; Renal function assessed by calculated creatinine clearance ≥ 30ml/min by Cockcroft-Gault formula; Total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST/SGOT) and alanine transaminase (ALT/SGPT) ≤ 2.5 x ULN; Alkaline phosphatase <2.5 x ULN
* Disease free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
* All study participants must be registered into the mandatory REMS® program, and be willing and able to comply with the requirements of REMS®.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid (ASA) may use warfarin or low molecular weight heparin).

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
* Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Evidence of laboratory Tumor Lysis Syndrome (TLS) by Cairo-Bishop Definition. Patients may be enrolled upon correction of electrolyte abnormalities.
* Use of any other experimental drug or therapy within 28 days of baseline
* Known hypersensitivity to thalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide
* Concurrent use of other anti-cancer agents or treatments
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV)
* Positive serology for hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive and HBsAb negative, a HB DNA test will be performed and if positive the patient will be excluded. Note: If HBcAb positive and HBsAb positive, which is indicative of a past infection, the patient can be included. Patients who are seropositive because of hepatitis B virus vaccine are eligible. Consult with a physician experienced in care & management of subjects with hepatitis B to manage/treat subjects who are anti-HBc positive.
* Positive serology for hepatitis C (HC) defined as a positive test for hepatitis C antibody (HCAb), in which case reflexively perform a HC recombinant immunoblot assay (RIBA) on the same sample to confirm the result
* Patients who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment) are ineligible.
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months prior to randomization, congestive heart failure [New York Heart Association (NYHA) III-IV], and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-03-30 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2024-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Bello, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immunotherapy
Started | 45
Completed | 44
Not Completed | 1
Not completed — Withdrew - received stem cell transplant | 1

BASELINE CHARACTERISTICS:
Arm/Group | Immunotherapy
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 44
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (CR)
Description: Number of participants with complete response, the disappearance of all signs of cancer in response to treatment.
Time Frame: 3 Months
Population: number of evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Immunotherapy
Number analyzed (Participants) | 44
Participants | 1

2. Primary Outcome: Number of Participants With Partial Response (PR)
Description: The primary endpoint for this trial is the combined complete and partial response rate to the protocol therapy at 3 months, which is also the end of Cycle 3. The objective response (CR+PR) rate will be summarized using both a point estimate and its exact confidence interval based on the binomial distribution.
Time Frame: 3 Months
Measure: Number; unit: participants
Arm/Group | Immunotherapy
Number analyzed (Participants) | 44
participants | 33

3. Secondary Outcome: Rate of Progression/Relapse Free Survival (PFS)
Description: Progression-free survival (PFS), defined as the time from study entry to disease progression, relapse or death due to any cause, whichever is earlier.
Time Frame: Up to 56 months
Population: evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Immunotherapy
Number analyzed (Participants) | 24
months | 54.4 [2.9 to 77.6]

4. Secondary Outcome: Number of Participants With Overall Survival (OS)
Description: Overall survival will be summarized with the Kaplan-Meier curve.
Time Frame: 36 Months
Population: evaluable participants
Measure: Number; unit: participants
Arm/Group | Immunotherapy
Number analyzed (Participants) | 24
participants | 24

ADVERSE EVENTS:
Time Frame: Adverse events collected from day 1 up to 30 days after cycle 12, 3 years and 6 months
Arm/Group | Immunotherapy
All-Cause Mortality (participants affected / at risk) | 6/45
Serious Adverse Events (participants affected / at risk) | 11/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy (N=45)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Fever (General disorders) | 2 (4)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy (N=45)
Fatigue (General disorders) | 22 (40)
Pain (General disorders) | 18 (30)
Infusion related reaction (General disorders) | 16 (20)
Edema limbs (General disorders) | 14 (24)
Fever (General disorders) | 13 (17)
Chills (General disorders) | 12 (15)
Flu like symptoms (General disorders) | 11 (14)
General disorders & administration site conditions-Other (General disorders) | 7 (8)
Irritability (General disorders) | 4 (4)
Non-cardiac chest pain (General disorders) | 3 (4)
Edema face (General disorders) | 2 (2)
Edema trunk (General disorders) | 2 (7)
Gait disturbance (General disorders) | 2 (2)
Injection site reaction (General disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Localized edema (General disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 37 (274)
White blood cell decreased (Investigations) | 29 (130)
Platelet count decreased (Investigations) | 16 (46)
Investigations -Other (Investigations) | 11 (22)
Alanine aminotransferase increased (Investigations) | 10 (24)
Aspartate aminotransferase increased (Investigations) | 8 (13)
Lymphocycte count decreased (Investigations) | 6 (7)
Creatinine increased (Investigations) | 5 (6)
Weight loss (Investigations) | 4 (6)
Alkaline phosphatase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (3)
Weight gain (Investigations) | 2 (2)
Lymphocyte count increased (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Metabolism and nutrition disorders -Other (Metabolism and nutrition disorders) | 34 (108)
Hyperkalemia (Metabolism and nutrition disorders) | 16 (29)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (21)
Anorexia (Metabolism and nutrition disorders) | 12 (15)
Hypermagnesemia (Metabolism and nutrition disorders) | 7 (8)
Hyperuricemia (Metabolism and nutrition disorders) | 6 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (18)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (9)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (11)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 4 (11)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 24 (48)
Constipation (Gastrointestinal disorders) | 20 (33)
Nausea (Gastrointestinal disorders) | 20 (33)
Dyspepsia (Gastrointestinal disorders) | 10 (15)
Abdominal Pain (Gastrointestinal disorders) | 9 (10)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 9 (12)
Dry mouth (Gastrointestinal disorders) | 6 (10)
Dysphagia (Gastrointestinal disorders) | 5 (5)
Flatulence (Gastrointestinal disorders) | 4 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Oral pain (Gastrointestinal disorders) | 4 (4)
Bloating (Gastrointestinal disorders) | 3 (4)
Stomach pain (Gastrointestinal disorders) | 3 (3)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (4)
Hemorrhoids (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 22 (34)
Headache (Nervous system disorders) | 19 (32)
Movements involuntary (Nervous system disorders) | 17 (26)
Dizziness (Nervous system disorders) | 15 (23)
Paresthesia (Nervous system disorders) | 13 (27)
Dysgeusia (Nervous system disorders) | 9 (14)
Concentration impairment (Nervous system disorders) | 7 (7)
Memory impairment (Nervous system disorders) | 7 (8)
Nervous system disorders - Other (Nervous system disorders) | 6 (7)
Tremor (Nervous system disorders) | 6 (8)
Akathisia (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Dyphasia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (5)
Sinus pain (Nervous system disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 19 (30)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 16 (25)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 15 (20)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (25)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (18)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 6 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (23)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (19)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 14 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (20)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (13)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 8 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 17 (23)
Sinusitis (Infections and infestations) | 14 (16)
Infections and infestations - Other (Infections and infestations) | 9 (9)
Urinary tract infection (Infections and infestations) | 5 (6)
Rash pustular (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Bronchial infection (Infections and infestations) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (2)
Mucosal infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 31 (53)
Anxiety (Psychiatric disorders) | 9 (14)
Depression (Psychiatric disorders) | 7 (8)
Psychiatric disorders - Other (Psychiatric disorders) | 7 (9)
Agitation (Psychiatric disorders) | 4 (5)
Confusion (Psychiatric disorders) | 2 (3)
Euphoria (Psychiatric disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (4)
Hypertension (Vascular disorders) | 19 (26)
Flushing (Vascular disorders) | 6 (9)
Hot flashes (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 5 (8)
Thromboembolic event (Vascular disorders) | 2 (2)
Lymphedema (Vascular disorders) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (1)
Vascular disorders - Other (Vascular disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 12 (20)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 7 (9)
Leukocytosis (Blood and lymphatic system disorders) | 5 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Lymph node pain (Blood and lymphatic system disorders) | 3 (5)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Eye disorders - Other (Eye disorders) | 15 (18)
Blurred vision (Eye disorders) | 7 (7)
Dry eye (Eye disorders) | 5 (6)
Watering eyes (Eye disorders) | 2 (2)
Cataract (Eye disorders) | 1 (2)
Floaters (Eye disorders) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (19)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Renal and urinary disorders - Other (Renal and urinary disorders) | 7 (11)
Urinary frequency (Renal and urinary disorders) | 5 (5)
Urinary retention (Renal and urinary disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (3)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (3)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 15 (26)
Cardiac disorders - Other (Cardiac disorders) | 8 (11)
Sinus bradycardia (Cardiac disorders) | 3 (6)
Sinus tachycardia (Cardiac disorders) | 3 (4)
Cardiac arrest (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 6 (7)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 3 (6)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT01496976/Prot_SAP_000.pdf